CLINICAL TRIAL: NCT05871177
Title: Pilot Study to Evaluate the Safety and Efficacy of 3.2% High (HHA) and Low (LHA) Molecular Weight Hyaluronic Acid Sodium Salt [32 Mg (HHA) + 32 Mg (LHA) / 2 Ml] for Intralesional Penile Injection in Peyronie's Disease
Brief Title: Safety and Efficacy of Intralesional HiLow Hyaluronic Acid in the Treatment of Peyronie's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPPPRVL/01-20
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm, multicentric, pilot clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HiLow hyaluronic acid sodium salt for intralesional penile injection (Experimental): Five intralesional injections of HiLow hyaluronic acid sodium salt will be administered in total to men affected by PD every two weeks (for a total period of 2.5 months). Patients will be then followed-up for 3 months.
  The following visits are scheduled:
  Day 0: basal visit Day 15: injection n.1 Day 30: injection n.2 Day 45: injection n.3 Day 60: injection n.4 Day 75: injection n.5 Day 180: end of follow up
  Interventions: Device: Pre-filled syringe of HiLow Hyaluronic Acid Sodium Salt

INTERVENTIONS:
Device: Pre-filled syringe of HiLow Hyaluronic Acid Sodium Salt — The medical device consists of a pre-filled syringe containing 3.2% Hyaluronic Acid Sodium Salt with high and low molecular weight [32 mg (HHA) + 32 mg (LHA) / 2 ml]

SUMMARY:
Prospective, open-label, single-arm, multicentric, pilot clinical study to confirm the safety of HiLow hyaluronic acid sodium salt for intralesional penile injection in patients affected by PD.

DETAILED DESCRIPTION:
Prospective, open-label, single-arm, multicentric, pilot clinical study to confirm the safety of HiLow hyaluronic acid sodium salt for intralesional penile injection in patients affected by PD.

Fourty patients aged 18-75 and affected by PD in the acute phase will be enrolled in the study.

The primary endpoint is the incidence of adverse events with causal relationship during the 2.5 months of active treatment and during follow-up.

The scondary endpoint is the overall improvement of the clinical condition by evaluation of the patient's global improvement (PGI-I scale), the amelioration in the degree of the curvature of the penis and the amelioration in the length of the penis after the induction of penile erection.

ELIGIBILITY:
Inclusion Criteria:

* basal degree of penile curvature not less than 30°
* preserved erection
* documented absence of coagulation defects (at least one examination of coagulation factors within the 3 months prior to the start of the study)
* written informed consent

Exclusion Criteria:

* presence of hourglass deformity
* presence of calcified plaques
* congenital curvature of the penis
* previous penile surgery
* concomitant oral treatment for IPP
* ongoing intralesional therapy or in the 3 months prior to the start of the study
* use of any traction device
* clinically stable disease
* history of symptomatic disease > 12 months
* known hypersensitivity or allergies to the components of the product
* any other clinical condition judged by the investigator not to be compatible with the participation in this study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From Day 0 to Day 180
  Evaluation of the safety of the treatment by measurement of the incidence of adverse events

SECONDARY OUTCOMES:
Patient's global impression of improvement | Day 75, Day 180
  Evaluation of patient's global impression of improvement by Patient Global Impression of Improvement (PGI-I) scale with a score from 1 (very much better) to 7 (very much worse).
Penile curvature | Day 0, Day 75, Day 180
  Evaluation of the amelioration in the degree of curvature of the penis measured using a goniometer
Penile length | Day 0, Day 75, Day 180
  Evaluation of the amelioration in the length of the penis after the induction of penile erection

CONTACTS AND LOCATIONS:
Overall Officials: Franco Gadda, MD, Principal Investigator — Fondazione IRCSS Cà Granda Ospedale Maggiore Policlinico
Locations (3):
- Italy (3):
  - U.O.C. Urologia, Azienda Ospedaliero Universitaria Mater Domini di Catanzaro, Catanzaro
  - Azienda Ospedaliero Universitaria delle Marche, Macerata
  - Fondazione IRCSS Cà Granda Ospedale Maggiore Policlinico, Milan